CLINICAL TRIAL: NCT05189236
Title: The Effect of Cold Steam Application on Body Temperature in Fever Management in Children with Febrile Neutropenia
Brief Title: Fever Management in Children with Febrile Neutropenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assist. Prof., Acibadem University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-Clinical Trials 2021/18
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2023-07

CONDITIONS: Fever
Keywords: Cold Steam; Body Temperature; Fever
MeSH Terms: conditions — Fever | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Only Algorithm of Febrile Neutropenia Management) (Other): The algorithm of febril neutropenia management is used to treat children who are followed up at the paediatric oncology service, where the study will be conducted, due to febrile neutropenia. The control group will consist of children who have been treated using this algorithm (only the Algorithm of Febrile Neutropenia Management).
  Interventions: Procedure: Control Group (Only Algorithm of Febrile Neutropenia Management)
- Experimental Group (Algorithm of Febrile Neutropenia Management+Cold Steam) (Experimental): The experimental group will consist of the children who will be applied to cold steam in addition to this algorithm (Algorithm of Febrile Neutropenia Management + cold steam application).
  Interventions: Procedure: Experimental Group (Algorithm of Febrile Neutropenia Management+Cold Steam)

INTERVENTIONS:
Procedure: Control Group (Only Algorithm of Febrile Neutropenia Management) — Common Procedure Steps
  1. The child is admitted to the unit and evaluated.
  2. The objective of the study is explained to the children and children's parents, and their consent is obtained after they have read and signed the informed consent form.
  3. The inclusion and exclusion criteria are evaluated.
  4. The group of the child to be included in the study is determined in accordance with the randomization order.
  5. The first section of the patient information and follow-up form is filled out.
  6. The algorithm of Febrile Neutropenia Management is applied. The room temperature is kept constant at 21-24 degrees.
  Procedure Steps for Control Group:
  1. Common procedure steps are followed.
  2. The body temperature of the child are recorded in the second section of the Patient Information and Follow-up Form until the fever is kept under control (until the discharge criteria are met, - 72 hours without fever and the culture result is negative).
  Arms: Control Group (Only Algorithm of Febrile Neutropenia Management)
Procedure: Experimental Group (Algorithm of Febrile Neutropenia Management+Cold Steam) — Procedure Steps for Experiment Group:
  1. Common procedure steps are followed.
  2. Cold steam is continuously applied until the fever is kept under control (until the discharge criteria are met, - 72 hours without fever and the culture result is negative).
  3. The body temperature of the child are recorded in the second section of the Patient Information and Follow-up Form from the time the patient is admitted until the fever is kept under control (until the discharge criteria are met, - 72 hours without fever and the culture result is negative).
  Arms: Experimental Group (Algorithm of Febrile Neutropenia Management+Cold Steam)

SUMMARY:
The aim of this study is to determine the effect of the cold steam application on body temperature in combination with the treatment algorithm in fever management in children with febrile neutropenia.

DETAILED DESCRIPTION:
Fever and neutropenia are common side effects of the myelosuppressive chemotherapy paediatric oncology patients undergo. This is one of the most prevalent causes of non-elective hospitalizations in patients in the population, accounting for 19% of patient applications. The fever that develops with neutropenia can result in significant complications, including brain damage, seizures and death. Therefore, it is critical to follow up patients at risk for signs and symptoms of infection, such as fever, chills or sweating, and to ensure effective fever management.

This research was designed to be conducted as a randomised controlled experiment study until the entire sample group identified in the Paediatric Oncology Service was reached. The algorithm of neutropenia management is used to treat children who are followed up at the paediatric oncology service, where the study will be conducted, due to febrile neutropenia. The control group will consist of children who have been treated using this algorithm (only the algorithm); whereas, the experimental group will consist of the children who will be applied to cold stream in addition to this algorithm (the algorithm + cold steam application). The body temperature values of patients in the experimental and control groups will be compared (from baseline to discharge (average 3 days)).

Cold Steam Application A nebulizer is positioned in the room, and the hose end, through which the steam is released, is supplied to the ambient air and operated in continuous mode during the cold steam application.

An Atom Sanilizer 30 ultrasonic nebulizer will be used to supply cold steam to every patient. The steam capacity of the device is 2.5 ml./min., the output power is 30 W.

The nebulizer will be used solely in the patient's room from the time the patient is admitted until his temperature is stabilised. During the private use period, the machine will not be exchanged between patients. During patient use, the device is cleaned with alcohol-based rapid surface disinfectant once a day. If another patient needs it, another device in the clinic will be utilized. The unit and the hospital already have a sufficient number of devices. After the patients' usage of the nebulizer is ended, the appliance is cleaned by using an alcohol-based rapid surface disinfectant, and the accessories are sterilized with a medium-level disinfectant in the Central Sterilization Unit.

During the practice of cold steam, if the body temperature falls within the usual range (axillary 36-37 0C, tympanic 36.5-37.7 0C), the practice will be discontinued and possible hypothermia will be avoided.

Procedures to follow in the development of hypothermia;

* ABC is evaluated.
* He is monitorised.

  -If there is no pulse, Advanced Life Support begins.
* A warm ambient is provided.
* He is warmed up with a blanket.

ELIGIBILITY:
Inclusion Criteria:

* The children and/or children's parents have agreed to participate in the study and have signed the informed consent form and
* Who are from the age of one month to eighteen years old,
* Children treated for febrile neutropenia
* Have a stable clinical condition will be included in the study

Exclusion Criteria:

* The children who have received a treatment protocol other than the algorithm of neutropenia management will be excluded from the study.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Body temperature | From baseline to discharge (average 3 days)
  The body temperature values of patients in the experimental and control groups will be compared (from baseline to discharge (average 3 days). Body temperature measurement will be evaluated as axillary.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assist Prof, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem Health Group Maslak Hospital, Istanbul, Maslak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson K, Bradford N, Edwards R, Nicholson J, Lockwood L, Clark JE. Improving management of fever in neutropenic children with cancer across multiple sites. Eur J Cancer Care (Engl). 2021 May;30(3):e13413. doi: 10.1111/ecc.13413. Epub 2021 Jan 28. PMID 33511731
- [Background] Green C, Krafft H, Guyatt G, Martin D. Symptomatic fever management in children: A systematic review of national and international guidelines. PLoS One. 2021 Jun 17;16(6):e0245815. doi: 10.1371/journal.pone.0245815. eCollection 2021. PMID 34138848
- [Background] Jung TH, Rho JH, Hwang JH, Lee JH, Cha SC, Woo SC. The effect of the humidifier on sore throat and cough after thyroidectomy. Korean J Anesthesiol. 2011 Dec;61(6):470-4. doi: 10.4097/kjae.2011.61.6.470. Epub 2011 Dec 20. PMID 22220223
- [Background] Lehrnbecher T. Treatment of fever in neutropenia in pediatric oncology patients. Curr Opin Pediatr. 2019 Feb;31(1):35-40. doi: 10.1097/MOP.0000000000000708. PMID 30461508
- [Background] Paolino J, Mariani J, Lucas A, Rupon J, Weinstein H, Abrams A, Friedmann A. Outcomes of a clinical pathway for primary outpatient management of pediatric patients with low-risk febrile neutropenia. Pediatr Blood Cancer. 2019 Jul;66(7):e27679. doi: 10.1002/pbc.27679. Epub 2019 Mar 27. PMID 30916887
- [Background] Taplitz RA, Kennedy EB, Flowers CR. Outpatient Management of Fever and Neutropenia in Adults Treated for Malignancy: American Society of Clinical Oncology and Infectious Diseases Society of America Clinical Practice Guideline Update Summary. J Oncol Pract. 2018 Apr;14(4):250-255. doi: 10.1200/JOP.18.00016. Epub 2018 Mar 8. No abstract available. PMID 29517953